CLINICAL TRIAL: NCT03968198
Title: Autologous Transplantation of Adipose Tissue Derived Mesenchymal Stroma/Stem Cells (ASC) in Patients With Critical Limb Ischemia.
Brief Title: Administration of Adipose-derived Stem Cells (ASC) in Patient With Critical Limb Ischemia.
Acronym: ACellDREAM2
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: organizational difficulties for the collection of adipose tissue and for the supply of the experimental drug
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/14/7441
Record Dates: First submitted 2019-05-14; First posted 2019-05-30 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Critical Limb Ischemia and Peripheral Artery Disease
Keywords: Cell therapy; ASC autologous; CLI; PAD; No option
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASC (Adipose-derived Stem/Stroma Cells) (Experimental): Patients administrated with autologous ASC in their ischemic inferiors limbs
  Interventions: Drug: Autologous ASC (for Adipose-derived Stem/Stroma Cell)

INTERVENTIONS:
Drug: Autologous ASC (for Adipose-derived Stem/Stroma Cell) — After adipose tissue aspiration (liposuction) by an authorized person, ASCs were isolated and cultured during 14±2 days by the French Blood Establishment. Then, patients receive intramuscular injections of ASCs.

SUMMARY:
Different types of stem cells have recently been studied in clinical trial on ischemic disease of the heart and muscular arteries. Adipose derived stem cell, have shown in vitro and in vivo models a stronger potential of success in recovering from ischemic disease and oxygenation of the tissues. The investigators already shown in a phase I study, that adipose derived mesenchymal cells injected in patients with critical limb ischemia and no option for revascularization, had a very good tolerance and interesting effects on skin oxygenation and healing.

The aim of the present clinical trial is to confirm the efficacy autologous transplantation of adipose tissue derived mesenchymal cells in patients with critical limb ischemia with poor options or no option for revascularization.

DETAILED DESCRIPTION:
Lower limbs arteries are a frequent localization of atheroma in elderly people (15-20% after 70 years). The most severe stage of the disease, critical limb ischemia (CLI), defined clinically by the presence of rest pain or ischemic ulcer, has a dramatic prognosis at 12 months, with 30% of the patients alive with an amputation, 20% mortality and only 20% of patients with a resolved disease, independently from the treatment. The only validated treatment for this disease is revascularization by endovascular procedures or open surgery. Patients with no option or poor option (high risk) for revascularization have the worst prognosis.

Current research is focusing on the development of cell-based therapies using different sources of stem cells which can provide revascularization and oxygenation of the tissues. A specific form of stem cells, called Adipose-derived Stem/Stroma Cells (ASC), has shown promise for recovering from ischemic disease like critical limb ischemia (CLI) in preclinical trial and trial in phase I. This study will confirm the efficacy autologous transplantation of adipose tissue derived mesenchymal cells in patients with critical limb ischemia with poor options or no option for revascularization.

This study is a phase II, prospective, multicentric, open trial and no comparative. A maximum of 43 patients will be included in two-stage to receive 90*106 intramuscular injection of ASC. Patients will be followed-up for 6 months.

The primary endpoint is the number of patients alive without major amputation and without critical limb ischemia (defined as the presence of rest pain or ischemic ulcer and ankle pressures less than 70 mmHg or toe systolic pressure less than 50 mmHg or TcPO2 of less than 30 mmHg, at six month).

The secondary endpoints are to evaluate:

* the number of new vessels in the treated limb by standardized angiographic magnetic resonance
* the blood flow by laser Doppler, transcutaneous pressure of oxygen (TcPO2), ankle pressure
* the percentage reduction of wound surface and percentage of complete ulcer healing
* the pain reduction by standardized evaluation (visual scale and drug consumption)
* the percentage of wound infection and irritative dermatitis (expected adverse events)
* interleukin-1, interleukin-2, interleukin-4, interleukin-6, interleukin-10, interleukin-12, Tumor Necrosis Factor alpha (TNFα)measurements in blood samples
* Mesenchymal stem cells MSC trophic factors and immune- modulators (Hepatocyte growth factor (HGF), Vascular Endothelial Growth Factor (VEGF), indoleamine 2, 3-dioxygenase (IDO), Human Leucocyte Antigen G (HLA-G)) in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old,
* Rest pain or ischemic ulcers /gangrene of the lower limb, present for at least 15 days, requiring analgesic absorption, with ankle pressures less than 70 mmHg or toe systolic pressure less than 50 mmHg or TcPO2 of less than 30 mmHg

Patient with persistent CLI after revascularization will be included if :

1. they have severe cardiac, respiratory or renal disease who are at increased risk of complication from surgery or anesthesia, e.g. moderately severe or severe heart failure (NYHA class III or IV), severe or very severe Chronic Obstructive Pulmonary disease or severe renal disease (creatinine clearance <30 mL/minute).

   OR
2. there is no option for endovascular or open surgery revascularization ; or poor option (defined by: need for an infra-popliteal by-pass without the availability of autologous great saphenous vein, need for use of great saphenous vein <3 mm in diameter for tibial level bypass based on venous duplex ultrasound, or calcified or small (<2 mm) distal target vessel, or open wound on the receiving site or infrapopliteal PAD)

   * Patients who signed the informed consent,
   * Patient affiliated to a social security system

Exclusion Criteria:

* History of cancer
* Need of a major amputation (amputation at or above the ankle) within 2 weeks,
* Ulcers with exposure of tendons, osteomyelitis, or clinically uncontrolled infection,
* TcPO2 <10 mmHg at rest and < 30 mmHg sitting with legs dependent (very poor vascular reserve),
* Patient under judicial protection,
* Pregnant women,
* Women of childbearing age without effective contraception.
* Refusal of the patient to participate in the study,
* Positive HIV-1 or 2, Human T Leukemia virus (HTLV)-1 or 2, Hepatite B Virus (HBV) (except vaccine profile), Syphilis (except inactive disease), or Hepatite C Virus (HCV)
* Patients necessitating drugs with inhibitory or stimulatory effect on the growth and multiplication of cells or drugs with immunosuppressive effect: Cyclosporine, Mycophenolate mofetil, Azathioprine, Tacrolimus (systemic), Anthracyclines, Neupogen or equivalent, Etanercept, Interferons, Corticoids at anti-inflammatory doses.
* No possibility of adipose tissue harvest and cell injection in the leg
* Another clinical trial participation (except non interventional studies),
* Patient under judicial protection,
* Pregnant and breastfeeding women,
* Women of childbearing age without effective contraception,
* Lack in understanding the nature and aims of the study and/or difficulties in communication with the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Number of patients alive without major amputation | Between 1 and 6 months
  Evaluation of the presence of rest pain or ischemic ulcer and ankle pressures less than 70 mmHg or toe systolic pressure less than 50 mmHg or TcPO2 of less than 30 mmHg, at six month.
Number of patients alive without critical limb ischemia | Between 1 and 6 months
  Evaluation of the presence of rest pain or ischemic ulcer and ankle pressures less than 70 mmHg or toe systolic pressure less than 50 mmHg or TcPO2 of less than 30 mmHg, at six month.

SECONDARY OUTCOMES:
New vessels | Between 1 and 6 months
  Blind evaluation of the number of new vessels in the treated limb by standardized angiographic magnetic resonance
Blood flow | Between 1 and 6 months
  Evaluation of the blood flow by laser Doppler, transcutaneous pressure of oxygen (TcPO2), ankle pressure.
Wound surface reduction | Between 1 and 6 months
  Percentage reduction of wound surface (standardized layer measurement).
Ulcer healing | Between 1 and 6 months
  Evaluation of percentage of complete ulcer healing.
Pain reduction | Between 1 and 6 months
  Evaluation of pain reduction by standardized evaluation (visual scale and drug consumption).
  The visual scale is in a form of plastic ruler and measures the intensity of pain on a scale ranging from 0 (no pain) to 10 (maximum pain).
Wound infection | Between 1 and 6 months
  Percentage of wound infection and irritative dermatitis (expected adverse events)
Immuno measures in blood sample | Between 1 and 6 months
  interleukin-1, interleukin-2, interleukin-4, interleukin-6, interleukin-10, interleukin-12, Tumor Necrosis Factor alpha (TNFα), will be measured out in blood samples.
Immuno measures in vitro | Between 1 and 6 months
  Mesenchymal stem cells (MSC) trophic factors and immune- modulators (Hepatocyte growth factor (HGF), Vascular Endothelial Growth Factor (VEGF), indoleamine 2, 3-dioxygenase (IDO), Human Leucocyte Antigen G (HLA-G)) will be studied in vitro.

CONTACTS AND LOCATIONS:
Overall Officials: BURA-RIVIERE Alessandra, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Rangueil Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dubsky M, Husakova J, Sojakova D, Fejfarova V, Jude EB. Cell Therapy of Severe Ischemia in People with Diabetic Foot Ulcers-Do We Have Enough Evidence? Mol Diagn Ther. 2023 Nov;27(6):673-683. doi: 10.1007/s40291-023-00667-w. Epub 2023 Sep 22. PMID 37740111